CLINICAL TRIAL: NCT02131272
Title: A 26-week Open Label, Randomised, 2-armed, Parallel Group, Multi-centre Trial Investigating Efficacy and Safety of Insulin Detemir Versus Insulin Neutral Protamine Hagedorn in Combination With the Maximum Tolerated Dose of Metformin and Diet/Exercise on Glycaemic Control in Children and Adolescents With Type 2 Diabetes Insufficiently Controlled on the Maximum Tolerated Dose of Metformin ± Other Oral Antidiabetic Drug(s) ± Basal Insulin
Brief Title: A Trial Investigating the Efficacy and Safety of Insulin Detemir Versus Insulin NPH in Combination With Metformin and Diet/Exercise in Children and Adolescents With Type 2 Diabetes Insufficiently Controlled on Metformin With or Without Other Oral Antidiabetic Drug(s) With or Without Basal Insulin
Acronym: iDEAt2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-4093; 2013-005500-33 (EudraCT Number); U1111-1151-4056 (Other: WHO); 2015-1316 (Registry Identifier: REec)
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Results first posted 2017-09-01 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin detemir and diet/exercise (Experimental): Current OADs i.e. metformin or other OADs are continued unchanged
  Interventions: Drug: Insulin NPH; Behavioral: Diet/exercise
- Insulin NPH and diet/exercise (Active Comparator): Current OADs i.e. metformin or other OADs are continued unchanged
  Interventions: Drug: Insulin detemir; Behavioral: Diet/exercise

INTERVENTIONS:
Drug: Insulin detemir — Administered subcutaneously (s.c., under the skin) once or twice daily. The subjects' pre-trial OAD's i.e. metformin treatment should continue unchanged during the treatment period.
  Arms: Insulin NPH and diet/exercise
Drug: Insulin NPH — Administered subcutaneously (s.c., under the skin) once or twice daily. The subjects' pre-trial OADs i.e. metformin treatment should continue unchanged during the treatment period.
  Arms: Insulin detemir and diet/exercise
Behavioral: Diet/exercise — Intervention will be performed through family based changes in eating and activity behaviours.

SUMMARY:
This trial is conducted globally. The aim of the trial is to investigate the efficacy and safety of insulin detemir versus insulin Neutral Protamine Hagedorn (NPH) in combination with the maximum tolerated dose of metformin and diet/exercise on glycaemic control in children and adolescents with type 2 diabetes insufficiently controlled on the maximum tolerated dose of metformin with or without other oral antidiabetic drug(s) with or without basal insulin.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from the subject or a legally acceptable representative (LAR) and child assent from the subject obtained before any trial-related activities.Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male or female, above or equal to 10 years and below or equal to 17 years at the time of signing informed consent/assent
* Diagnosis of type 2 diabetes mellitus at least 3 months prior to screening
* Treated with the maximum tolerated stable dose of metformin for at least 3 months prior to screening or have documented complete metformin intolerance
* HbA1c (glycosylated haemoglobin) above or equal to 7.0% and below or equal to 10.5% (above or equal to 53 mmol/mol and below or equal to 91 mmol/mol) at screening

Exclusion Criteria:

* Maturity onset diabetes of the young (MODY)
* Fasting C-peptide at screening below 0.6 ng/mL
* Impaired liver function defined as alanine aminotransferase (ALT) above or equal to 2.5 times upper normal limit
* Known proliferative retinopathy or maculopathy requiring acute treatment as judged by the investigator
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 3 months before the day of screening

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2014-06-11 (Actual); Primary Completion 2016-06-14 (Actual); Study Completion 2016-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (73):
- United States (22):
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Tallahassee, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Reisterstown, Maryland
  - Novo Nordisk Investigational Site, Silver Spring, Maryland
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Buffalo, New York
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Toledo, Ohio
  - Novo Nordisk Investigational Site, Hershey, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Providence, Rhode Island
  - Novo Nordisk Investigational Site, Columbia, South Carolina
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Edinburg, Texas
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Novo Nordisk Investigational Site, CABA, Argentina
- Brazil (3):
  - Novo Nordisk Investigational Site, Aparecida de Goiânia, Goiás
  - Novo Nordisk Investigational Site, Porto Alegre, Rio Grande do Sul
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
- Novo Nordisk Investigational Site, Zagreb, Croatia
- Egypt (2):
  - Novo Nordisk Investigational Site, Alexandria
  - Novo Nordisk Investigational Site, Cairo
- Germany (2):
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Neuwied
- Greece (2):
  - Novo Nordisk Investigational Site, Goudi/ Athens
  - Novo Nordisk Investigational Site, Thessaloniki
- Hungary (2):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Miskolc
- India (5):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
- Israel (2):
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Haifa
- Italy (2):
  - Novo Nordisk Investigational Site, Ancona
  - Novo Nordisk Investigational Site, Florence
- Lebanon (3):
  - Novo Nordisk Investigational Site, Beirut
  - Novo Nordisk Investigational Site, Hazmiyeh
  - Novo Nordisk Investigational Site, Lebanon - Beirut
- Malaysia (4):
  - Novo Nordisk Investigational Site, Kota Kinabalu
  - Novo Nordisk Investigational Site, Kuala Lumpur
  - Novo Nordisk Investigational Site, Seremban
  - Novo Nordisk Investigational Site, Seri Manjung
- Novo Nordisk Investigational Site, Puebla City, Mexico
- Morocco (4):
  - Novo Nordisk Investigational Site, Casablanca
  - Novo Nordisk Investigational Site, Fes
  - Novo Nordisk Investigational Site, Marrakesh
  - Novo Nordisk Investigational Site, Rabat
- Novo Nordisk Investigational Site, Wroclaw, Poland
- Novo Nordisk Investigational Site, Lisbon, Portugal
- Russia (3):
  - Novo Nordisk Investigational Site, Izhevsk
  - Novo Nordisk Investigational Site, Stavropol
  - Novo Nordisk Investigational Site, Tomsk
- Novo Nordisk Investigational Site, Niš, Serbia
- South Africa (3):
  - Novo Nordisk Investigational Site, Lenasia, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Observatory, Western Cape
- Novo Nordisk Investigational Site, Seoul, South Korea
- Novo Nordisk Investigational Site, Esplugues Llobregat(Barcelona), Spain
- Taiwan (2):
  - Novo Nordisk Investigational Site, Taichung
  - Novo Nordisk Investigational Site, Taoyuan District
- Turkey (Türkiye) (4):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Kayseri

REFERENCES:
- [Result] Wheeler MD, Barrientos-Perez M, Lo FS, Liang B, Lunsford A, Thorisdottir O, Zuckerman-Levin N. A 26-week, randomized trial of insulin detemir versus NPH insulin in children and adolescents with type 2 diabetes (iDEAt2). Eur J Pediatr. 2018 Oct;177(10):1497-1503. doi: 10.1007/s00431-018-3205-z. Epub 2018 Jul 16. PMID 30014302
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The following 12 countries screened subjects (no. of sites that randomised subjects within parentheses): Brazil (1), Germany (1), India (3), Israel (1), South Korea (1), Malaysia (3), Mexico (1), Russian Federation (1) Taiwan (3), Turkey (3), United States (6), Hungary (0). A total of 24 sites in 11 countries randomised subjects to treatment.
Pre-assignment Details: Subjects continued treatment with metformin on their pre-study dose(s) throughout the trial.
Groups:
- Insulin Detemir + Metformin + Diet/Exercise: Subjects were treated with insulin detemir 100 U/mL administered subcutaneously in the thigh region once or twice daily for a period of 26 weeks. For insulin naïve subjects, insulin detemir was initiated at a dose of 0.1-0.2 U/kg with a maximum dose of 10 U at the investigators discretion. Subjects who were already on basal insulin were switched to insulin detemir unit-to-unit once or twice daily, depending on previous injection frequency. Subjects were dosed according to individual requirements during the trial period. All subjects continued treatment with metformin on their pre-study dose(s) throughout the trial. The diet/exercise intervention was performed through changes in eating and activity behaviours.
- Insulin NPH + Metformin + Diet/Exercise: Subjects were treated with NPH 100 IU/mL administered subcutaneously in the thigh region once or twice daily for a period of 26 weeks. For insulin naïve subjects, insulin NPH was initiated at a dose of 0.1-0.2 U/kg with a maximum dose of 10 U at the investigators discretion. Subjects who were already on basal insulin were switched to insulin NPH unit-to-unit once or twice daily, depending on previous injection frequency. Subjects were dosed according to individual requirements during the trial period. All subjects continued treatment with metformin on their pre-study dose(s) throughout the trial. The diet/exercise intervention was performed through changes in eating and activity behaviours.
Period: Overall Study
Arm/Group | Insulin Detemir + Metformin + Diet/Exercise | Insulin NPH + Metformin + Diet/Exercise
Started | 20 | 22
Completed | 19 | 20
Not Completed | 1 | 2
Not completed — Withdrawal by parent | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Withdrawal Criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Detemir + Metformin + Diet/Exercise | Insulin NPH + Metformin + Diet/Exercise | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.0 (2.1) | 15.0 (2.2) | 15.0 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 8 | 7 | 15
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.72 (0.86) | 8.95 (1.05) | 8.84 (0.96)
Body weight standard deviation score [Mean (Standard Deviation); unit: standard deviation score] — In order to reduce the variability in body weight measurements, standard deviation scores (SDS) were calculated. SDS for weight was derived by comparing the actual measurements with standard growth charts for the United States. Standard values provided by the standard growth charts according to the subject's sex and age at the time of the measurement were used to calculate the SDS.
  standard deviation score | 1.532 (0.685) | 1.260 (0.835) | 1.390 (0.771)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Glycosylated Haemoglobin)
Description: Estimated mean change in HbA1c (glycosylated haemoglobin) from baseline to week 26.
Time Frame: week 0, week 26
Population: Full analysis set included all the randomised subjects.
Measure: Least Squares Mean (Standard Error); unit: Percentage of glycosylated haemoglobin
Arm/Group | Insulin Detemir + Metformin + Diet/Exercise | Insulin NPH + Metformin + Diet/Exercise
Number analyzed (Participants) | 20 | 22
Percentage of glycosylated haemoglobin | -0.64 (0.32) | -0.81 (0.31)
Statistical Analysis 1: Comparison: Insulin Detemir + Metformin + Diet/Exercise vs Insulin NPH + Metformin + Diet/Exercise; HbA1c measurements were analysed with a mixed model for repeated measurements with an unstructured covariance matrix. The model included treatment, visit, age group, prior antidiabetic therapy and interaction between prior antidiabetic therapy and age group as fixed factors and the HbA1c baseline value as covariate. Interactions between visit and all factors and covariates were also included in the model; Test type: Non-Inferiority or Equivalence — Non-inferiority was considered fulfilled if the upper bound of the two-sided 95% confidence interval for the difference between detemir and NPH was below or equal to 0.4%. The sample size was set to ensure 80% power for the full analysis set (FAS). However, efficacy conclusions cannot be drawn from the analysis due to low number of subjects included in the trial; p = 0.3075, Mixed Models Analysis — p value is reported for 1 sided test; Least squares mean difference = 0.17, 95% CI 2-sided [-0.74 to 1.09]

2. Secondary Outcome: Change in Body Weight Standard Deviation Score (SDS)
Description: Change in body weight standard deviation score (SDS) from baseline to week 26. In order to reduce the variability in body weight measurements, SDS were calculated. SDS for weight was derived by comparing the actual measurements with standard growth charts for the United States. Standard values provided by the standard growth charts according to the subject's sex and age at the time of the measurement were used to calculate the SDS.
Time Frame: week 0, week 26
Population: Full analysis set included all the randomised subjects.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | Insulin Detemir + Metformin + Diet/Exercise | Insulin NPH + Metformin + Diet/Exercise
Number analyzed (Participants) | 20 | 22
standard deviation score | 0.006 (0.192) | 0.098 (0.139)

3. Secondary Outcome: Proportion of Subjects Achieving HbA1c Below 7.0%, Who Have Not Experienced Any Treatment Emergent Severe Hypoglycaemic Episodes Within the Last 14 Weeks of Treatment.
Description: Proportion of subjects achieving HbA1c <7.0% is presented as percentage of subjects achieving HbA1c <7.0%, who have not experienced any treatment emergent severe hypoglycaemic episodes (an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) within the last 14 weeks of treatment.
Time Frame: At week 26
Population: Full analysis set included all the randomised subjects. Only subjects who have been exposed for a minimum of 14 weeks contributed to the analysis (20 subjects in the Insulin detemir + metformin + diet/exercise arm and 21 subjects in the Insulin NPH + metformin + diet/exercise arm).
Measure: Number; unit: Percentage of subjects
Arm/Group | Insulin Detemir + Metformin + Diet/Exercise | Insulin NPH + Metformin + Diet/Exercise
Number analyzed (Participants) | 20 | 21
Percentage of subjects | 25.0 | 33.3

4. Secondary Outcome: Proportion of Subjects Achieving HbA1c Below 7.5%, Who Have Not Experienced Any Treatment Emergent Severe Hypoglycaemic Episodes Within the Last 14 Weeks of Treatment
Description: Proportion of subjects achieving HbA1c below 7.5% is presented as percentage of subjects achieving HbA1c <7.5%, who have not experienced any treatment emergent severe hypoglycaemic episodes (an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) within the last 14 weeks of treatment.
Time Frame: At week 26
Population: as for outcome 3
Measure: Number; unit: Percentage of subjects
Arm/Group | Insulin Detemir + Metformin + Diet/Exercise | Insulin NPH + Metformin + Diet/Exercise
Number analyzed (Participants) | 20 | 21
Percentage of subjects | 30.0 | 38.1

5. Secondary Outcome: Total Number of Treatment Emergent Nocturnal (23:00-06:59) Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemic Episodes
Description: The total number of blood glucose confirmed symptomatic nocturnal (time of onset between 23:00 and 06.59 both inclusive) severe (an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or blood glucose confirmed symptomatic hypoglycaemic episodes (plasma glucose value <3.1 mmol/L [56 mg/dL] with symptoms consistent with hypoglycaemia) experienced by the subjects during the trial.
Time Frame: Weeks 0 - 26
Population: Safety analysis set included all subjects receiving at least one dose of randomised treatment.
Measure: Number; unit: Number of episodes
Arm/Group | Insulin Detemir + Metformin + Diet/Exercise | Insulin NPH + Metformin + Diet/Exercise
Number analyzed (Participants) | 20 | 22
Number of episodes
  Severe | 0 | 0
  Blood glucose confirmed symptomatic | 0 | 1

6. Secondary Outcome: Total Number of Treatment Emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: Total number of treatment emergent severe (an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or blood glucose confirmed symptomatic hypoglycaemic episodes (plasma glucose value <3.1 mmol/L [56 mg/dL] with symptoms consistent with hypoglycaemia) experienced by the subjects during the trial.
Time Frame: Weeks 0 - 26
Population: Safety analysis set included all subjects receiving at least one dose of randomised treatment.
Measure: Number; unit: Number of episodes
Arm/Group | Insulin Detemir + Metformin + Diet/Exercise | Insulin NPH + Metformin + Diet/Exercise
Number analyzed (Participants) | 20 | 22
Number of episodes
  Severe | 0 | 0
  Blood glucose confirmed symptomatic | 4 | 12

7. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: The total number of treatment emergent adverse events (the onset of the adverse event is on or after the first day of trial product administration, and no later than 7 days after the last day of trial product administration) reported during the 26 weeks of treatment.
Time Frame: weeks 0 - 26
Population: Safety analysis set included all subjects receiving at least one dose of randomised treatment.
Measure: Number; unit: Number of events
Arm/Group | Insulin Detemir + Metformin + Diet/Exercise | Insulin NPH + Metformin + Diet/Exercise
Number analyzed (Participants) | 20 | 22
Number of events | 30 | 41

ADVERSE EVENTS:
Time Frame: Adverse events from the first trial-related activity (week -2) after the subject and/or his/her legally acceptable representative has signed the informed consent until the end of the trial (week 26).
Description: Safety analysis set included all subjects receiving at least one dose of randomised treatment.
  A treatment emergent adverse event was defined as an event that had the onset date on or after the first day of trial product administration, and no later than 7 days after the last day of trial product administration.
Arm/Group | Insulin Detemir + Metformin + Diet/Exercise | Insulin NPH + Metformin + Diet/Exercise
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/22
Other Adverse Events (participants affected / at risk) | 8/20 | 9/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir + Metformin + Diet/Exercise (N=20) | Insulin NPH + Metformin + Diet/Exercise (N=22)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir + Metformin + Diet/Exercise (N=20) | Insulin NPH + Metformin + Diet/Exercise (N=22)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 1 (4)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (3)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was terminated earlier than planned due to a very slow recruitment rate. Based on the low number of subjects, the conclusions should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.